CLINICAL TRIAL: NCT06626542
Title: EFFECT OF INTRA-SESSION EXERCISE MODES SEQUENCE ON VENTRICULAR FUNCTION IN PATIENTS WITH CHRONIC HEART FAILUIRE
Brief Title: Effect of Intra-session Exercise Modes Sequence on Ventricular Function in Patients With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasser Mostafa Mohamed Elhamamsy, Yasser Mostafa Mohamed El-hamamsy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004786
Record Dates: First submitted 2024-06-02; First posted 2024-10-04 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sequence of aerobic cardiovascular training (CVT) then resistance training (RT) exercises (Experimental)
  Interventions: Other: resistance and aerobic training exercises
- sequence of resistance training (RT) then aerobic cardiovascular training (CVT) exercises (Experimental)
  Interventions: Other: resistance and aerobic training exercises
- control group routine treatment programme only (Other)
  Interventions: Other: resistance and aerobic training exercises

INTERVENTIONS:
Other: resistance and aerobic training exercises — resistance and aerobic training exercises
  Other Names: cardiac rehabilitation

SUMMARY:
The aim of this study was to investigate the effect of intra-session exercise modes sequence on ventricular function in patients with chronic heart failure.

DETAILED DESCRIPTION:
Sixty male patients with chronic heart failure will be recruited in this study from National Heart Institute Giza, Egypt. Their ages will be ranged from 55 to 65 years old and they will be randomly divided into three groups as following:

1. Study group (A) includes 20 patients who will receive intra-session exercise modes sequence of aerobic cardiovascular training (CVT) then resistance training (RT) exercises in addition to routine treatment programme.
2. Study group (B) includes 20 patients who will receive intra-session exercise modes sequence of resistance training (RT) then aerobic cardiovascular training (CVT) exercises in addition to routine treatment programme.
3. Control group (C) includes 20 patients who will receive routine treatment programme only.

The exercise training programme for both study groups A and B will be applied once per day, three times per week for 12 consecutive weeks.

Inclusion criteria:

All participated patients will be:

* Male patients with chronic heart failure and ages from 55 to 65 years old.
* Class II and class III heart failure according to NYHA classification.
* HFrEF category with LVEF <40% as documented by echocardiogram within <6 months.
* Receiving the same medical treatment programme for at least 3 months.
* Having a close level of functional capacity assessed by 6 minute walking test.

Exclusion criteria:

Patients who meet one of the following criteria will be excluded:

* Uncontrolled atrial fibrillation.
* Diabetes mellitus.
* Myocardial infarction or recurrent angina within <3 months.
* Patients with chronic chest diseases.
* Severe stenotic valvular disease.
* Clinically significant peripheral vascular disease.
* Exercise-induced angina, ST segment changes or exercise induce AV block.
* Patients with chronic renal failure.
* Any cognitive impairment that interferes with prescribed exercise procedures.
* Musculoskeletal or neurological limitation to physical exercise.

RESEARCH ETHICS

The protocol of this study will be approved by the ethics committee of scientific research at the Faculty of Physical Therapy, Cairo University. The study procedure will be explained in details for every patient before the initial assessment. All patients will be informed about the purpose, nature, and potential risks of the study, and a written informed consent will be obtained before participation in the study. The participants' right confidentiality will be observed strictly.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with chronic heart failure and ages from 55 to 65 years old.

  * Class II and class III heart failure according to NYHA classification.
  * HFrEF category with LVEF <40% as documented by echocardiogram within <6 months.
  * Receiving the same medical treatment programme for at least 3 months.
  * Having a close level of functional capacity assessed by 6 minute walking test

Exclusion Criteria:

* • Uncontrolled atrial fibrillation.

  * Diabetes mellitus.
  * Myocardial infarction or recurrent angina within <3 months.
  * Patients with chronic chest diseases.
  * Severe stenotic valvular disease.
  * Clinically significant peripheral vascular disease.
  * Exercise-induced angina, ST segment changes or exercise induce AV block.
  * Patients with chronic renal failure.
  * Any cognitive impairment that interferes with prescribed exercise procedures.
  * Musculoskeletal or neurological limitation to physical exercise.

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — males only
Enrollment: 60 (Actual)
Dates: Start 2023-09-03 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 12 weeks
  left ventricular ejection fraction is measured by using echocardiography it is measured in percentage %

SECONDARY OUTCOMES:
The Minnesota living with heart failure questionnaire (MLWHFQ) | 12 weeks
  calculate minnasota living with heart failure questionnaire score 21 item MLHFQ uses a 6-point scale where 0 = no, 1= very little and 5= very much
Cardiorespiratory fitness 6 minute walk test | 12 weeks
  after the test we calculate the distance patient walked in meters and we use this distance to evaluate the cardiopulmonary fitness
Vo2 Max | 12 week
  by using distance from the 6MWT in meters we can calculate the vo2 max using specific equation
Blood pressure | 12 weeks
  blood pressure systolic by using the sphygmomanometer palpatory method - diastolic by using the auscultatory method by sphygmomanometer and stethoscope
Rate of pressure product | 12 week
  rate pressure product will be calculated by this equation : patient heart rate * systolic blood pressure / 1000

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Institute, Giza, Agouza Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided